CLINICAL TRIAL: NCT06125665
Title: Impacts of Aminophylline on Perioperative Lung Mechanics in COPD Morbidly Obese Patients Undergoing Laparoscopic Bariatric Surgery: A Prospective Randomized Double Blinded Trial
Brief Title: Aminophylline on Perioperative Lung Mechanics in COPD Morbidly Obese Patients Undergoing Laparoscopic Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Soliman Ramadan Ahmed Naser, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR361/9/23
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Aminophylline; Chronic Obstructive Pulmonary Disease; Obese; Laparoscopic Bariatric Surgery; Dexmedetomidine; Lung Mechanics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aminophylline-Dexmedetomidine Group (Experimental): 10 minutes after endotracheal intubation, patients will receive IV bolus of dexmedetomidine 0.5 microgm/kg Lean body weight (LBW) over 15 min, followed immediately by intravenous infusion at 0.2 microgm /kg LBW/h and IV bolus of aminophylline of 5 mg/kg based on the ideal body weight (IBW) over 30 min, followed immediately by intravenous infusion at 0.6 mg/kg IBW/h. The study solutions will be diluted in 50 ml normal saline.
  Interventions: Drug: Aminophylline-Dexmedetomidine
- Dexmedetomidine (Active Comparator): 10 minutes after endotracheal intubation, patients will receive IV bolus of dexmedetomidine 0.5 microgm/kg LBW over 15 min, followed immediately by intravenous infusion at 0.2 microgm /kg LBW/h. The study solutions will be diluted in 50 ml normal saline.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Aminophylline-Dexmedetomidine — 10 minutes after endotracheal intubation, patients will receive intravenous (IV) bolus of dexmedetomidine 0.5 microgm/kg Lean body weight (LBW) over 15 min, followed immediately by intravenous infusion at 0.2 microgm /kg LBW/h and IV bolus of aminophylline of 5 mg/kg based on the ideal body weight (IBW) over 30 min, followed immediately by intravenous infusion at 0.6 mg/kg IBW/h. The study solutions will be diluted in 50 ml normal saline.
  Arms: Aminophylline-Dexmedetomidine Group
Drug: Dexmedetomidine — 10 minutes after endotracheal intubation, patients will receive intravenous (IV) bolus of dexmedetomidine 0.5 microgm/kg Lean body weight (LBW) over 15 min, followed immediately by intravenous infusion at 0.2 microgm /kg LBW/h. The study solutions will be diluted in 50 ml normal saline.
  Arms: Dexmedetomidine

SUMMARY:
The aim of this study is to evaluate the usefulness of adding aminophylline to dexmedetomidine intravenous infusion intraoperatively on oxygenation and lung mechanics in chronic obstructive pulmonary disease (COPD) morbidly obese patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
Bariatric surgery is considered the most effective treatment for patients suffering from morbid obesity, as it results in maintained loss of weight and clear impact on the comorbidities related to obesity. However, despite the advantages of anesthesia, it can have detrimental effects on the recovery of obese patients who have a high prevalence of respiratory conditions and sleep disorders.

Obesity is usually related to other respiratory diseases such as asthma, chronic obstructive pulmonary disease (COPD). According to a meta-analysis encompassing more than 300,000 adult patients, obesity and asthma were interlinked, and as BMI increased, a higher risk of asthma was noticed.

The use of dexmedetomidine infusion in morbid obese patients was assessed by many clinical trials. They revealed that the use of dexmedetomidine has the same analgesic effect as the use of fentanyl with greater hemodynamic stability obtained with the use of dexmedetomidine. Dexmedetomidine has the advantage of having no respiratory depressant effect. Also, it has an amnestic effect. Dexmedetomidine does not affect the sleep pattern and maintains the airway patency.

Aminophylline is a compound of theophylline with ethylenediamine and most common uses in the airway obstruction such as asthma and COPD. primarily for its bronchodilating and central nervous stimulating effects. However, emprical evidence suggests that aminophylline, as an adenosine antagonist, can improve the recovery time from general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 60 years.
* Patients scheduled for laparoscopic bariatric surgery not exceeding three hours under general anesthesia.
* American Society of Anesthesiologists (ASA) class II to III.
* Patients who had no previous abdominal surgery.
* Patients with a body mass index (BMI) greater than 40 kg/m2and suffered obstructive lung disease diagnosed by pulmonary function tests (; forced vital capacity (FEV1\FVC) < 70%).
* Patients who are psychologically normal.

Exclusion Criteria:

* Patients who refuse to participate.
* Those with arrhythmia or receiving anti-arrhythmic medications.
* Those with significant coexisting diseases (e.g. kidney, heart, liver).
* Those with known allergy to any of allocated drugs.
* Those with excessive intraoperative blood loss more than allowable amount to every patient.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Static lung compliance | Up to 90 minutes after the beginning of the drug infusion.
  Static lung compliance will be calculated as: tidal volume/ [plateau pressure - Positive end-expiratory pressure (PEEP)] at 5 minutes after endotracheal intubation (baseline), 30 and 90 minutes after the beginning of the drug infusion.

SECONDARY OUTCOMES:
Dynamic lung compliance | Up to 90 minutes after the beginning of the drug infusion.
  Dynamic lung compliance will be calculated as: tidal volume/ [peak airway pressure - Positive end-expiratory pressure (PEEP)] at 5 minutes after endotracheal intubation (baseline), 30 and 90 minutes after the beginning of the drug infusion.
Intraoperative oxygenation | Up to 90 minutes after the beginning of the drug infusion.
  Intraoperative oxygenation will be measured at 5 minutes after endotracheal intubation (baseline), 30 and 90 minutes after the beginning of the drug infusion determined by (S/F ratio: SPO2/ FiO2).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.